CLINICAL TRIAL: NCT05863884
Title: RADx-UP- Impact of Community Health Worker Home Deployment on COVID-19 Vaccine Confidence and Uptake
Brief Title: RADx-UP- Impact of Community Health Worker Deployment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1854646
Record Dates: First submitted 2022-12-02; First posted 2023-05-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; COVID-19; Community Health Workers; Health Behavior; Health Knowledge, Attitudes, Practice
Keywords: diabetes; COVID-19; rural communities; rural health center; rural population; community health workers
MeSH Terms: conditions — Diabetes Mellitus; COVID-19; Health Behavior; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CHW Intervention (Other): A six week CHW home-visit behavioral intervention examining changes in diabetes outcomes.
  Interventions: Behavioral: Impact of Community Health Worker Home Deployment on COVID-19 Vaccine Confidence and Uptake

INTERVENTIONS:
Behavioral: Impact of Community Health Worker Home Deployment on COVID-19 Vaccine Confidence and Uptake — CHWs will conduct home visits to provide diabetes and COVID-19 health education based on the participant's needs, interests, and clinical health assessment results. All adults in the household will be invited to participate in the health education discussions. At each visit, the CHW will use diabetes management and COVID-19 educational materials to facilitate and inform discussions. CHWs will also make available at-home COVID-19 testing kits with instructions for the patient and their household family members. The discussion of COVID-19 beliefs, perceptions, and related behaviors will be raised during a later visit, i.e., after rapport and trust has been established and if it has not been raised by the participants during the earlier visits. In addition, CHWs will help schedule vaccination and healthcare appointments upon participant's interest.

SUMMARY:
The proposed project will implement and evaluate a brief Community Health Worker (CHW) intervention through the Albany Area Primary Health Care, a rural Federally Qualified Health Center (FQHC). The primary goal of this study is to maximize effective outreach, education, and communication through CHWs in order to facilitate improved COVID-19 vaccine confidence and uptake in underserved and vulnerable communities. CHWs will be deployed to the homes of adults with increased risk of morbidity and mortality (i.e., African Americans or Latinos with uncontrolled diabetes or prediabetes, age <50 years, and non-COVID-19 vaccinated) in order to educate them about diabetes, COVID-19 and related vaccines. Health assessments, including blood glucose measurement, will be conducted on the indexed patient and offered to all other adult family members in the household (i.e., "bubble"). Adults with Type 2 diabetes likely live in households with other adults who have or are at increased risk for diabetes (i.e., prediabetes and obesity).1 It is expected that they will also share similar COVID-19 exposure risk. The specific aims are to: 1) Evaluate a community-driven education program to increase and enhance COVID-19 vaccine confidence and uptake in individuals with uncontrolled diabetes and their families (i.e., their "bubble") and 2) Evaluate a community-driven education program to improve diabetes self-management behaviors and related outcomes (e.g., blood glucose) in individuals with uncontrolled diabetes in rural, Southwest Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between18 and 50 years
* Self-identify as African American/Black or Latino
* English speaking
* Have received care for uncontrolled diabetes (HbA1c > 9%) or prediabetes diagnosis within one of the AAPHC 27 community sites
* Unvaccinated for Phase 1 (vaccinated for Phase 2)

Exclusion Criteria:

* Not meeting the Inclusion Criteria
* Enrolled in the parent RADx-UP Project PEACH study
* Unable or unwilling to provide informed consent to participate in the study (ie: incarcerated individuals and children)
* Individuals with a terminal cancer diagnosis, have chronic kidney disease (stage 4-5), pregnant women, and people with severe psychological disorders (i.e., dementia,suicide ideation)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Level | 6 weeks
  Change in HbA1c level from using clinical assessment parameters from week 1 to week 6.

SECONDARY OUTCOMES:
Diabetes Self-Management Score | 6 weeks
  Change in overall diabetes self-management score using diabetes self-management questionnaire from week 1 to week 6.

OTHER OUTCOMES:
COVID-19 Vaccination Confidence and Uptake | 6 weeks
  Change in COVID-19 vaccination status and confidence using diabetes self-management questionnaire from week 1 to week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Rakale C Quarells, PhD, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Albany Area Primary Health Care, Albany, Georgia, United States

IPD SHARING:
Plan to Share IPD: No